CLINICAL TRIAL: NCT03401125
Title: Retrospective Study of the Risk Factors for Allo-immunization in Sickle Cell Disease
Brief Title: Risk Factors for Allo-immunization in Sickle Cell Disease
Status: Withdrawn | Type: Observational
Why Stopped: Results already published by another team
Sponsor: Hanane EL KENZ (Other)
Responsible Party: Sponsor-Investigator, Hanane EL KENZ, Head of Blood Bank, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-RETRO-ALLO
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Allo-immunization
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle cell disease patients (SS genotype): Sickle cell disease patients with a SS genotype having an history of blood transfusions within the CHU Brugmann and the Queen Fabiola Children's Hospitals.
  Interventions: Other: Medical file data collection

INTERVENTIONS:
Other: Medical file data collection — The information described in the 'outcome measures' section will be collected from the medical files of the patients.

SUMMARY:
Sickle cell patients have a high prevalence of alloimmunization. This high rate of alloimmunization can be partially explained by the existence of an antigenic difference between the predominantly Caucasian donor population and the sickle cell patients of African origin. Genetic and environmental risk factors have also been described.

The main risk factors that have been shown in retrospective or cross-sectional studies are some HLA alleles, the age of the patient, the number of leukocyte-depleted erythrocyte concentrates (CED) transfused, the number of transfusion episodes, the age of the CEDs, the existence of an inflammatory event at the time of transfusion and the presence of anti-erythrocyte autoantibodies.There is also evidence of an impaired TH response but the underlying immunological mechanism is not fully understood.

The aim of this study is to study the prevalence and the risk factors for anti-erythrocyte alloimmunization in pediatric and adult patients with Sickle Cell Disease (with a SS genotype) who are being followed at Queen Fabiola University Children's Hospital (HUDERF) and at the CHU Brugmann Hospital. The identification of risk factors would allow the investigators to improve, or at least adapt, their transfusion policy to certain clinical or immuno-haematological situations.

ELIGIBILITY:
Inclusion Criteria:

- Sickle cell disease patients (HbSS genotype) with a history of blood transfusions within the CHU Brugmann and the Queen Fabiola University Hospitals.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sickle cell disease patients (HbSS genotype) with a history of blood transfusion within the CHU Brugmann and the Queen Fabiola University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Date of birth | january 2013-december 2017
  Date of birth
Sex | january 2013-december 2017
  Sex
Blood group | january 2013-december 2017
  Blood group
Extended phenotype | january 2013-december 2017
  Sickle cell disease extended phenotype
Antibodies | january 2013-december 2017
  Presence/absence of irregular anti-erythrocytes antibodies (RAI)
Number of blood transfusions | january 2013-december 2017
  Number of blood transfusions
Number of blood transfusions | From birth till the first positive RAI test (up to 50 years)
  Number of blood transfusions
Auto antibodies | january 2013-december 2017
  Presence/absence of auto anti-erythrocytes antibodies (RAI)
Pathology | january 2013-december 2017
  Medical issue causing the patient to be included in a chronic blood transfusion program
Duration of the chronic transfusion program | january 2013-december 2017
  Duration of the chronic transfusion program

CONTACTS AND LOCATIONS:
Overall Officials: Marie Deleers, Ph Biol, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - HUDERF, Brussels

IPD SHARING:
Plan to Share IPD: No